CLINICAL TRIAL: NCT05920122
Title: A Randomized Control Trial of Chlorhexidine Gluconate Aqueous Solution vs Chlorhexidine Gluconate With Isopropyl Alcohol Skin Preparations for Prevention of Cesarean Section Wound Infections
Brief Title: Aqueous vs Alcohol Chlorhexidine Skin Preparation for Prevention of Cesarean Section Wound Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hyagriv Simhan (Other)
Responsible Party: Sponsor-Investigator, Hyagriv Simhan, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY23030049
Record Dates: First submitted 2023-06-07; First posted 2023-06-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Surgical Site Infection; Cesarean Section; Infection
MeSH Terms: conditions — Surgical Wound Infection; Infections | interventions — chlorhexidine gluconate; Ethanol

STUDY DESIGN:
Intervention Model Description: Immediately prior to entering the operating room, participants will be randomly assigned in a 1:1 ratio to the CHG or CHG-IPA group. Groups will be stratified by laboring status defined as :
  1. Regular contractions with cervical dilation of 4 cm or more OR
  2. Documented cervical change of at least 1 cm of dilation or at least 50% effacement OR
  3. Rupture of membranes
Who Masked: Outcomes Assessor
Masking Description: The provider making the diagnosis of wound infection will be blinded to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2% Chlorhexidine gluconate with 70% alcohol (ChloraPrep) (Experimental): Including cases undergoing elective &non elective caesarean section. Patients will be prepared similarly using the appropriate number of 26mL Chloraprep sticks for their body surface area. The lever will be pinched to activate the ampoule and release the antiseptic. The solution will be given time to partially load in the sponge. The sponge will be pressed against the skin area where the incision is intended moving back and forth for 30 sec , then working up towards the upper edge of the surgical field and then working from below the incision sight to the upper thighs. The antiseptic will be given time to dry (3 min)
  Interventions: Drug: 2% Chlorhexidine gluconate with 70% alcohol
- 4% chlorhexidine gluconate (Hibiclens) (Experimental): Including cases undergoing elective & nonelective caesarean section. Patients will be scrubbed preoperative with an applicator that contain 4% chlorohexidine aqueous solution (3 consecutive applications) liberally over 2 minutes followed by drying with sterile towel. The area scrubbed will be the same as the chloraprep group.
  Interventions: Drug: 4% Chlorhexidine Gluconate aqueous solution

INTERVENTIONS:
Drug: 2% Chlorhexidine gluconate with 70% alcohol — Patients will be prepared similarly using the appropriate number of 26mL Chloraprep sticks for their body surface area. The lever will be pinched to activate the ampoule and release the antiseptic. The solution will be given time to partially load in the sponge. The sponge will be pressed against the skin area where the incision is intended moving back and forth for 30 sec , then working up towards the upper edge of the surgical field and then working from below the incision sight to the upper thighs. The antiseptic will be given time to dry (3 min)
  Other Names: ChloraPrep
  Arms: 2% Chlorhexidine gluconate with 70% alcohol (ChloraPrep)
Drug: 4% Chlorhexidine Gluconate aqueous solution — Patients will be scrubbed preoperative with an applicator that contain 4% chlorohexidine aqueous solution (3 consecutive applications) liberally over 2 minutes followed by drying with sterile towel. The area scrubbed will be the same as the chloraprep group.
  Other Names: Hibiclens
  Arms: 4% chlorhexidine gluconate (Hibiclens)

SUMMARY:
This will be a single-center randomized control trial comparing the efficacy of two different formulations of Chlorhexidine surgical skin preparation in preventing cesarean section wound infections. Participants will be randomized to either 4% Chlorhexidine Gluconate aqueous solution (CHG) or 2% Chlorhexidine with isopropyl alcohol (CHG-IPA) 70% to examine the risk of infectious morbidity in those undergoing cesarean delivery. There will also be a cost-effectiveness analysis of the two preoperative skin preparations.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing cesarean delivery at Magee Women's Hospital

Exclusion Criteria:

* Inability to obtain consent (language barrier, emergency cesarean section etc.)
* Allergy to chlorhexidine or alcohol
* Chorioamnionitis
* Emergency cesareans where cannot wait for chlorhexidine alcohol to dry
* bowel injury at time of cesarean section
* Women who are delivered at another institution and are transferred postpartum to Magees Women's Hospital

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1398 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Surgical site Infection | Within 30 days post cesarean
  Superficial or deep surgical-site infection within 30 days after cesarean delivery, on the basis of the National Healthcare Safety Network definitions of the Centers for Disease Control and Prevention.

SECONDARY OUTCOMES:
Number of Participants With Endometritis | Within 30 days post cesarean
Number of Participants with intrabdominal/pelvic abscess | Within 90 days post cesarean
Number of Participants with necrotizing fasciitis | Within 90 days post cesarean
Number of Participants with sepsis | Within 90 days post cesarean
  With wound/uterine infection as the source
Length of Hospital Stay | Within 90 days post cesarean
Number of Participants With Re-admissions or Office Visits for Wound-related Problems | Within 90 days post cesarean
Number of Participants with ICU admission for wound infectious complications | Within 90 days post cesarean
Number of Participants with Need for wound opening, exploration, or washout in the operating room | Within 90 days post cesarean
Number of Participants who needed wound vacuum | Within 90 days post cesarean
Number of Participants who needed home health | Within 90 days post cesarean
Number of patients who needed antibiotics | Within 90 days post cesarean
  will also collect route of antibiotic administration and duration of treatment to assist with cost analysis
Number of doses of antibiotic treatment | Within 90 days post cesarean
  for wound infection complications
Antibiotic regimens (medication names) used to treat infection | Within 90 days post cesarean
  for wound infection complications
Number of participants with positive culture from wound | Within 90 days post cesarean
The type of bacterial species isolated from wound infection cultures | Within 90 days post cesarean
Number of participants with hematoma | Within 90 days post cesarean
Number of participants with seroma | Within 30 days post cesarean
Number of Participants With Skin Irritation | within 48 hours from delivery
Number of Participants With Allergic Reaction | within 48 hours from delivery
Cost Savings | Within 90 days post cesarean
  costs (dollars) associated with a hospital stay, office visits and re-admissions for infection-related complications, ICU admission for infectious complications, wound exploration or washout in the operating room, wound vacuum use, home health, antibiotic prescriptions, and duration of treatment will be collected and used to calculate the cost of wound infection management. The cost difference between groups will be calculated to estimate cost savings.

CONTACTS AND LOCATIONS:
Overall Officials: Yaneve Fonge, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costantine MM, Rahman M, Ghulmiyah L, Byers BD, Longo M, Wen T, Hankins GD, Saade GR. Timing of perioperative antibiotics for cesarean delivery: a metaanalysis. Am J Obstet Gynecol. 2008 Sep;199(3):301.e1-6. doi: 10.1016/j.ajog.2008.06.077. PMID 18771991
- [Background] Saeed KB, Greene RA, Corcoran P, O'Neill SM. Incidence of surgical site infection following caesarean section: a systematic review and meta-analysis protocol. BMJ Open. 2017 Jan 11;7(1):e013037. doi: 10.1136/bmjopen-2016-013037. PMID 28077411
- [Background] Merkow RP, Ju MH, Chung JW, Hall BL, Cohen ME, Williams MV, Tsai TC, Ko CY, Bilimoria KY. Underlying reasons associated with hospital readmission following surgery in the United States. JAMA. 2015 Feb 3;313(5):483-95. doi: 10.1001/jama.2014.18614. PMID 25647204
- [Background] Zuarez-Easton S, Zafran N, Garmi G, Salim R. Postcesarean wound infection: prevalence, impact, prevention, and management challenges. Int J Womens Health. 2017 Feb 17;9:81-88. doi: 10.2147/IJWH.S98876. eCollection 2017. PMID 28255256
- [Background] Zimlichman E, Henderson D, Tamir O, Franz C, Song P, Yamin CK, Keohane C, Denham CR, Bates DW. Health care-associated infections: a meta-analysis of costs and financial impact on the US health care system. JAMA Intern Med. 2013 Dec 9-23;173(22):2039-46. doi: 10.1001/jamainternmed.2013.9763. PMID 23999949
- [Background] Darouiche RO, Wall MJ Jr, Itani KM, Otterson MF, Webb AL, Carrick MM, Miller HJ, Awad SS, Crosby CT, Mosier MC, Alsharif A, Berger DH. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. N Engl J Med. 2010 Jan 7;362(1):18-26. doi: 10.1056/NEJMoa0810988. PMID 20054046
- [Background] Ferrannini E, Santoro D, Manicardi V. The association of essential hypertension and diabetes. Compr Ther. 1989 Nov;15(11):51-8. PMID 2684484
- [Background] Springel EH, Wang XY, Sarfoh VM, Stetzer BP, Weight SA, Mercer BM. A randomized open-label controlled trial of chlorhexidine-alcohol vs povidone-iodine for cesarean antisepsis: the CAPICA trial. Am J Obstet Gynecol. 2017 Oct;217(4):463.e1-463.e8. doi: 10.1016/j.ajog.2017.05.060. Epub 2017 Jun 7. PMID 28599898
- [Background] Dumville JC, McFarlane E, Edwards P, Lipp A, Holmes A, Liu Z. Preoperative skin antiseptics for preventing surgical wound infections after clean surgery. Cochrane Database Syst Rev. 2015 Apr 21;2015(4):CD003949. doi: 10.1002/14651858.CD003949.pub4. PMID 25897764
- [Background] Caughey AB, Wood SL, Macones GA, Wrench IJ, Huang J, Norman M, Pettersson K, Fawcett WJ, Shalabi MM, Metcalfe A, Gramlich L, Nelson G, Wilson RD. Guidelines for intraoperative care in cesarean delivery: Enhanced Recovery After Surgery Society Recommendations (Part 2). Am J Obstet Gynecol. 2018 Dec;219(6):533-544. doi: 10.1016/j.ajog.2018.08.006. Epub 2018 Aug 15. PMID 30118692
- [Background] Maiwald M, Chan ES. Pitfalls in evidence assessment: the case of chlorhexidine and alcohol in skin antisepsis. J Antimicrob Chemother. 2014 Aug;69(8):2017-21. doi: 10.1093/jac/dku121. Epub 2014 Apr 28. PMID 24777898
- [Background] Hadiati DR, Hakimi M, Nurdiati DS, Masuzawa Y, da Silva Lopes K, Ota E. Skin preparation for preventing infection following caesarean section. Cochrane Database Syst Rev. 2020 Jun 25;6(6):CD007462. doi: 10.1002/14651858.CD007462.pub5. PMID 32580252
- [Background] Levin I, Amer-Alshiek J, Avni A, Lessing JB, Satel A, Almog B. Chlorhexidine and alcohol versus povidone-iodine for antisepsis in gynecological surgery. J Womens Health (Larchmt). 2011 Mar;20(3):321-4. doi: 10.1089/jwh.2010.2391. Epub 2011 Feb 16. PMID 21323582